CLINICAL TRIAL: NCT05707910
Title: A Phase I Study of the Efficacy and Safety of Therapeutic Immunological Agent for EBV-positive Advanced Malignant Tumors
Brief Title: Clinical Study of Therapeutic Immunological Agent for EBV-positive Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1389
Record Dates: First submitted 2023-01-09; First posted 2023-02-01 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Malignant Tumor
Keywords: EBV; tumor; immunotherapy
MeSH Terms: conditions — Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): EBV immunological agent administration on day 0,7,14,28 and 60 for subcutaneous injection.
  Interventions: Biological: EBV immunological agent

INTERVENTIONS:
Biological: EBV immunological agent — 2*10^7 and 5*10^7
  Other Names: Toripalimab 240mg

SUMMARY:
To evaluate the safety of therapeutic immunological agent against EBV-positive advanced malignancies, examining the incidence, type of occurrence, and severity of adverse events in relation to the agent tested, and initially exploring the effectiveness of the immunological agent.

DETAILED DESCRIPTION:
EBV (Epstein-Barr virus) is the first tumor-associated virus to be discovered, closely related to a variety of malignant tumors, including nasopharyngeal carcinoma (NPC), a variety of lymphomas, such as Hodgkin lymphoma (HL), non-Hodgkin lymphoma (NHL), Burkitt's lymphoma (BL) and partial EBV positive stomach cancer (EBV-associated Gastric Carcinomas, EBVaGC). Treatment of the above EBV+ tumors, surgery, radiotherapy and chemotherapy are still the main methods, immunotherapy for some patients has shown good efficacy, prolonging the patient's overall survival rate (Overall Survival, OS) and progression-free survival rate (Progression-Free-Survival, PFS), but the overall clinical efficacy needs to be further improved, and new treatment methods are urgently needed.

After tumor cells are infected with EBV virus, they will express a variety of EBV virus antigens, which these proteins can promote the transformation and proliferation of human cells, inhibit cell apoptosis and participate in the occurrence and development of tumors, which also become candidate targets for research of immunotherapy because of the strong antigenicity of viral antigens.

Therapeutic immunological agent was prepared which are naturally loaded with EBV antigens and present them to activate T cells and dendritic cells(DC) in vitro and significantly inhibit tumor growth in vivo. The agent also showed good safety. According to these findings suggest the therapeutic immunological agent provides a new idea for immunotherapy of EBV-related tumors.

The findings suggest that a number of patients with malignant tumors who failed EBV+ multi-line therapy, including nasopharyngeal cancer, NK/T lymphoma, and gastric cancer needed to be treated with new immunotherapy method to achieve better outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: ≥ 18 years old; ≤ 70 years old;
2. Patients with EBV-positive advanced malignant tumors after failure of second-line standard therapy (including PD-1 inhibitor therapy);
3. ECOG physical fitness score: 0~2 points;
4. Estimated survival ≥ 3 months;
5. The main organs have good function, that is, the relevant examination indicators within random 14 days meet the following requirements:

   1. Blood routine examination: hemoglobin ≥ 80 g/L (no blood transfusion within 14 days); Neutrophil count> 1.5×10^9/L; Platelet count≥ 80×10^9/L;
   2. Biochemical examination: total bilirubin ≤ 1.5× ULN (upper limit of normal); alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5×ULN; If liver metastases are present, ALT or AST ≤ 5×ULN; Endogenous creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula);
   3. Cardiac Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ 50%.
6. Sign the informed consent form;
7. Good compliance, family members agree to cooperate with survival follow-up.

Exclusion Criteria:

1. Participated in clinical trials of other drugs within 4 weeks;
2. The patient has a history of other tumors, unless it is cervical cancer in situ, treated cutaneous squamous cell carcinoma or bladder epithelial tumor or other malignant tumor that has received radical treatment (at least 5 years before enrollment)
3. Patients with uncontrolled cardiac clinical symptoms or diseases, such asheart failure above NYHA grade 2, unstable angina, myocardial infarction within 1 year, and clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
4. For female subjects: pregnant or lactating women.
5. The patient has active tuberculosis, bacterial or fungal infection; There is HIV infection with active HBV infection, HCV infection.
6. Those who have a history of psychotropic drug abuse and have mental disorders who cannot be remitted;
7. The subject has any active autoimmune disease or has a history of autoimmune disease (such as, but not limited to uveitis, enteritis, pituitary inflammation, nephritis, hyperthyroidism, hypothyroidism, Participants with vitiligo or who had complete remission of asthma in childhood and did not require any intervention in adulthood could be included; Participants in asthma requiring medical intervention with bronchodilators were not included).
8. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the patient's research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 12 months
  The primary endpoint was safety, with adverse events (AEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.
Objective response rate | up to 12 months
  ORR is defined as the percentage of patients who achieve a response, which can either be complete response (complete disappearance of lesions) or partial response (reduction in the sum of maximal tumor diameters by at least 30% or more)
Progress-Free Survival | up to 12 months
  PFS is defined as the time from the administration of the first dose to first disease
Overall Survival | up to 12 months
  OS is defined as the time from the administration of the first dose to death.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Downs-Canner SM, Meier J, Vincent BG, Serody JS. B Cell Function in the Tumor Microenvironment. Annu Rev Immunol. 2022 Apr 26;40:169-193. doi: 10.1146/annurev-immunol-101220-015603. Epub 2022 Jan 19. PMID 35044794
- [Background] Choi IK, Wang Z, Ke Q, Hong M, Paul DW Jr, Fernandes SM, Hu Z, Stevens J, Guleria I, Kim HJ, Cantor H, Wucherpfennig KW, Brown JR, Ritz J, Zhang B. Mechanism of EBV inducing anti-tumour immunity and its therapeutic use. Nature. 2021 Feb;590(7844):157-162. doi: 10.1038/s41586-020-03075-w. Epub 2020 Dec 23. PMID 33361812
- [Background] Klarquist J, Cross EW, Thompson SB, Willett B, Aldridge DL, Caffrey-Carr AK, Xu Z, Hunter CA, Getahun A, Kedl RM. B cells promote CD8 T cell primary and memory responses to subunit vaccines. Cell Rep. 2021 Aug 24;36(8):109591. doi: 10.1016/j.celrep.2021.109591. PMID 34433030
- [Background] Schriek P, Ching AC, Moily NS, Moffat J, Beattie L, Steiner TM, Hosking LM, Thurman JM, Holers VM, Ishido S, Lahoud MH, Caminschi I, Heath WR, Mintern JD, Villadangos JA. Marginal zone B cells acquire dendritic cell functions by trogocytosis. Science. 2022 Feb 11;375(6581):eabf7470. doi: 10.1126/science.abf7470. Epub 2022 Feb 11. PMID 35143312
- [Background] Rossetti RAM, Lorenzi NPC, Yokochi K, Rosa MBSF, Benevides L, Margarido PFR, Baracat EC, Carvalho JP, Villa LL, Lepique AP. B lymphocytes can be activated to act as antigen presenting cells to promote anti-tumor responses. PLoS One. 2018 Jul 5;13(7):e0199034. doi: 10.1371/journal.pone.0199034. eCollection 2018. PMID 29975708
- [Background] Laurell A, Lonnemark M, Brekkan E, Magnusson A, Tolf A, Wallgren AC, Andersson B, Adamson L, Kiessling R, Karlsson-Parra A. Intratumorally injected pro-inflammatory allogeneic dendritic cells as immune enhancers: a first-in-human study in unfavourable risk patients with metastatic renal cell carcinoma. J Immunother Cancer. 2017 Jun 20;5:52. doi: 10.1186/s40425-017-0255-0. eCollection 2017. PMID 28642820
- [Background] Eagles ME, Nassiri F, Badhiwala JH, Suppiah S, Almenawer SA, Zadeh G, Aldape KD. Dendritic cell vaccines for high-grade gliomas. Ther Clin Risk Manag. 2018 Jul 26;14:1299-1313. doi: 10.2147/TCRM.S135865. eCollection 2018. PMID 30100728
- [Background] Comoli P, Pedrazzoli P, Maccario R, Basso S, Carminati O, Labirio M, Schiavo R, Secondino S, Frasson C, Perotti C, Moroni M, Locatelli F, Siena S. Cell therapy of stage IV nasopharyngeal carcinoma with autologous Epstein-Barr virus-targeted cytotoxic T lymphocytes. J Clin Oncol. 2005 Dec 10;23(35):8942-9. doi: 10.1200/JCO.2005.02.6195. Epub 2005 Oct 3. PMID 16204009
- [Background] Bollard CM, Gottschalk S, Torrano V, Diouf O, Ku S, Hazrat Y, Carrum G, Ramos C, Fayad L, Shpall EJ, Pro B, Liu H, Wu MF, Lee D, Sheehan AM, Zu Y, Gee AP, Brenner MK, Heslop HE, Rooney CM. Sustained complete responses in patients with lymphoma receiving autologous cytotoxic T lymphocytes targeting Epstein-Barr virus latent membrane proteins. J Clin Oncol. 2014 Mar 10;32(8):798-808. doi: 10.1200/JCO.2013.51.5304. Epub 2013 Dec 16. PMID 24344220
- [Background] Lopez-Chavez A, Thomas A, Rajan A, Raffeld M, Morrow B, Kelly R, Carter CA, Guha U, Killian K, Lau CC, Abdullaev Z, Xi L, Pack S, Meltzer PS, Corless CL, Sandler A, Beadling C, Warrick A, Liewehr DJ, Steinberg SM, Berman A, Doyle A, Szabo E, Wang Y, Giaccone G. Molecular profiling and targeted therapy for advanced thoracic malignancies: a biomarker-derived, multiarm, multihistology phase II basket trial. J Clin Oncol. 2015 Mar 20;33(9):1000-7. doi: 10.1200/JCO.2014.58.2007. Epub 2015 Feb 9. PMID 25667274
- [Background] Cunanan KM, Gonen M, Shen R, Hyman DM, Riely GJ, Begg CB, Iasonos A. Basket Trials in Oncology: A Trade-Off Between Complexity and Efficiency. J Clin Oncol. 2017 Jan 20;35(3):271-273. doi: 10.1200/JCO.2016.69.9751. Epub 2016 Nov 28. No abstract available. PMID 27893325
- [Background] Cho J, Kang MS, Kim KM. Epstein-Barr Virus-Associated Gastric Carcinoma and Specific Features of the Accompanying Immune Response. J Gastric Cancer. 2016 Mar;16(1):1-7. doi: 10.5230/jgc.2016.16.1.1. Epub 2016 Mar 31. PMID 27104020
- [Background] Young LS, Dawson CW. Epstein-Barr virus and nasopharyngeal carcinoma. Chin J Cancer. 2014 Dec;33(12):581-90. doi: 10.5732/cjc.014.10197. Epub 2014 Nov 21. PMID 25418193
- [Background] Kanakry JA, Ambinder RF. EBV-related lymphomas: new approaches to treatment. Curr Treat Options Oncol. 2013 Jun;14(2):224-36. doi: 10.1007/s11864-013-0231-y. PMID 23549980
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Bekoz H, Karadurmus N, Paydas S, Turker A, Toptas T, Firatli Tuglular T, Sonmez M, Gulbas Z, Tekgunduz E, Kaya AH, Ozbalak M, Tastemir N, Kaynar L, Yildirim R, Karadogan I, Arat M, Pepedil Tanrikulu F, Ozkocaman V, Abali H, Turgut M, Kurt Yuksel M, Ozcan M, Dogu MH, Kabukcu Hacioglu S, Barista I, Demirkaya M, Koseoglu FD, Toprak SK, Yilmaz M, Demirkurek HC, Demirkol O, Ferhanoglu B. Nivolumab for relapsed or refractory Hodgkin lymphoma: real-life experience. Ann Oncol. 2017 Oct 1;28(10):2496-2502. doi: 10.1093/annonc/mdx341. PMID 28961828
- [Background] Kfoury M, Disdero V, Vicier C, Le Saux O, Gougis P, Sajous C, Vignot S. [Immune checkpoints inhibitors: Recent data from ASCO's meeting 2017 and perspectives]. Bull Cancer. 2018 Jul-Aug;105(7-8):686-695. doi: 10.1016/j.bulcan.2018.04.011. Epub 2018 Jun 20. French. PMID 29933886
- [Background] Holko P, Kawalec P. Economic evaluation of sipuleucel-T immunotherapy in castration-resistant prostate cancer. Expert Rev Anticancer Ther. 2014 Jan;14(1):63-73. doi: 10.1586/14737140.2014.856270. PMID 24224852
- [Background] Tanyi JL, Bobisse S, Ophir E, Tuyaerts S, Roberti A, Genolet R, Baumgartner P, Stevenson BJ, Iseli C, Dangaj D, Czerniecki B, Semilietof A, Racle J, Michel A, Xenarios I, Chiang C, Monos DS, Torigian DA, Nisenbaum HL, Michielin O, June CH, Levine BL, Powell DJ Jr, Gfeller D, Mick R, Dafni U, Zoete V, Harari A, Coukos G, Kandalaft LE. Personalized cancer vaccine effectively mobilizes antitumor T cell immunity in ovarian cancer. Sci Transl Med. 2018 Apr 11;10(436):eaao5931. doi: 10.1126/scitranslmed.aao5931. PMID 29643231
- [Background] Liau LM, Ashkan K, Tran DD, Campian JL, Trusheim JE, Cobbs CS, Heth JA, Salacz M, Taylor S, D'Andre SD, Iwamoto FM, Dropcho EJ, Moshel YA, Walter KA, Pillainayagam CP, Aiken R, Chaudhary R, Goldlust SA, Bota DA, Duic P, Grewal J, Elinzano H, Toms SA, Lillehei KO, Mikkelsen T, Walbert T, Abram SR, Brenner AJ, Brem S, Ewend MG, Khagi S, Portnow J, Kim LJ, Loudon WG, Thompson RC, Avigan DE, Fink KL, Geoffroy FJ, Lindhorst S, Lutzky J, Sloan AE, Schackert G, Krex D, Meisel HJ, Wu J, Davis RP, Duma C, Etame AB, Mathieu D, Kesari S, Piccioni D, Westphal M, Baskin DS, New PZ, Lacroix M, May SA, Pluard TJ, Tse V, Green RM, Villano JL, Pearlman M, Petrecca K, Schulder M, Taylor LP, Maida AE, Prins RM, Cloughesy TF, Mulholland P, Bosch ML. First results on survival from a large Phase 3 clinical trial of an autologous dendritic cell vaccine in newly diagnosed glioblastoma. J Transl Med. 2018 May 29;16(1):142. doi: 10.1186/s12967-018-1507-6. PMID 29843811
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949